CLINICAL TRIAL: NCT04656717
Title: Cost of Cancer Diagnosis Using Next-generation Sequencing Targeted Gene Panels in Routine Practice: a Nationwide French Study
Brief Title: Cost of Cancer Diagnosis Using Next-generation Sequencing Targeted Gene Panels in Routine Practice
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 29367707
Record Dates: First submitted 2019-05-26; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Cancer
Keywords: Next-generation sequencing (NGS); Cost; Cancer diagnosis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measure of the total cost of performing next-generation sequencing (NGS) — Resources consumed were collected for each laboratory using a standardized questionnaire. The production costs were calculated for the overall process and resources consumed for each step were identified.

SUMMARY:
The aim of this study was to measure the total cost of performing next-generation sequencing (NGS) in clinical practice in France, in both germline and somatic cancer genetics.

The study was performed on 15 French representative cancer molecular genetics laboratories performing NGS panels' tests. The production cost was estimated using a micro-costing method with resources consumed collected in situ in each laboratory from a healthcare provider perspective. A top-down methodology for specific post-sequencing steps was used.

Additional non-specific costs were also included and costs were detailed per step of the process.

ELIGIBILITY:
Inclusion Criteria:

* French genetics laboratories performing somatic and germline clinical NGS tests.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: French laboratories (7 somatic genetics and 8 germline oncogenetic) currently performing NGS.The laboratories were chosen because they performed cancer diagnostics nationwide and presented the full spectrum of clinical indications and technical solutions
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Overall production cost | through study completion, an average of 5 years
  The study is performed on 15 French representative cancer molecular genetics laboratories performing NGS panels' tests. The production cost is estimated using a micro-costing method with resources consumed collected in situ in each laboratory from a healthcare provider perspective. A top-down methodology for specific post-sequencing steps is used.

IPD SHARING:
Plan to Share IPD: No